CLINICAL TRIAL: NCT02419053
Title: Evaluating the Effect of Surgical Safety Checklists on Perioperative Complications in Children
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Institute for Clinical Evaluative Sciences (Other)
Responsible Party: Principal Investigator, James O'Leary, Staff Anesthesiologist, The Hospital for Sick Children
Other Study IDs: 1000046196
Record Dates: First submitted 2015-04-13; First posted 2015-04-17 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Intraoperative Complications; Postoperative Complications
Keywords: Surgical safety checklist; perioperative complications; pediatric
MeSH Terms: conditions — Intraoperative Complications; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre-checklist: Surgical interventions performed for children before the introduction of the surgical safety checklist in Ontario, from October 2008 to September 2009.
- Post-checklist: Surgical interventions performed for children after the introduction of the surgical safety checklist in Ontario, from October 2010 to September 2011.
  Interventions: Other: Surgical Safety Checklist

INTERVENTIONS:
Other: Surgical Safety Checklist — An Ontario hospital-wide introduction of a surgical safety checklist based on the WHO guidelines, as mandated by the Ontario Ministry of Health
  Groups: Post-checklist

SUMMARY:
The purpose of this study is to see if the surgical safety checklist is associated with a reduction in perioperative complications for children undergoing surgery in Ontario, Canada.

ELIGIBILITY:
Inclusion Criteria:

* Surgical admission, with a noncardiac surgical interventions
* Aged between >28 days and <18years on the day of the surgical intervention

Exclusion Criteria:

* Non-surgical admission
* Surgical interventions with <10 per group
* Cardio-thoracic and interventional cardiology procedures

Ages: 28 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Surgical interventions performed in Ontario for children
Sampling Method: Non-Probability Sample
Enrollment: 28772 (Actual)
Dates: Start 2008-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Perioperative complications | 30-days after surgery
  Composite outcome, complications included were death (all-causes), acute renal failure, cardiac arrest, complications of implants or grafts, decubitus ulcer, deep vein thrombosis, disruption of wound, electrolyte or acid-base abnormality, hemorrhage or hematoma, pulmonary embolism, pulmonary collapse or pneumonia, surgical site infection, sepsis, shock, stroke, and vascular graft failure

SECONDARY OUTCOMES:
Healthcare utilization - proportion of Emergency Room visits | 30-days after surgery
  Number of Emergency Room visits
Healthcare utilization - rate of unplanned return to the operating room | 30-days after surgery
  Unplanned return to the operating room
Healthcare utilization - length of hospital stay | 30-days after surgery
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: James D O'Leary, MBBCh, Principal Investigator — The Hospital for Sick Children, Toronto
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] O'Leary JD, Wijeysundera DN, Crawford MW. Effect of surgical safety checklists on pediatric surgical complications in Ontario. CMAJ. 2016 Jun 14;188(9):E191-E198. doi: 10.1503/cmaj.151333. Epub 2016 Mar 14. PMID 26976960